CLINICAL TRIAL: NCT04374721
Title: Clinical Study on Circadian Genes Dysregulation in Patients With Glucocorticoid Disorders
Acronym: CHROnOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Associate Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHROnOS
Record Dates: First submitted 2020-04-23; First posted 2020-05-05 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Cushing Syndrome; Adrenal Insufficiency; Cushing Disease; Addison Disease
Keywords: circadian rhythm; circadian genes; circadian clock; glucocorticoids; cortisol
MeSH Terms: conditions — Cushing Syndrome; Adrenal Insufficiency; Pituitary ACTH Hypersecretion; Addison Disease

STUDY DESIGN:
Intervention Model Description: patients will undergo circadian genes evaluation in peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Adrenal Insufficiency (Experimental): Patients with Adrenal Insufficiency established or newly diagnosed, under glucocorticoid replacement therapy.
  Interventions: Diagnostic Test: circadian gene expression evaluation
- Patients with Cushing's Syndrome (Experimental): patients with adrenocorticotropic hormone (ACTH)-dependent or ACTH-independent Cushing's Syndrome diagnosis during active disease (new diagnosis or recidivating) at enrollment.
  Interventions: Diagnostic Test: circadian gene expression evaluation
- Healthy Controls (Experimental): Age-, sex- and BMI- matched patients referring to our center for diagnostic procedures not affected by Adrenal Insufficiency or Cushing's Syndrome.
  Interventions: Diagnostic Test: circadian gene expression evaluation

INTERVENTIONS:
Diagnostic Test: circadian gene expression evaluation — patients and controls will undergo circadian gene expression (CLOCK, ARNTL) evaluation at baseline and after 1, 3 and 6 months

SUMMARY:
This is a multicentric, prospective, intervention study on circadian genes expression in peripheral blood mononuclear cells as biomarkers of circadian rhythm derangement in patients affected by alterations of endogenous glucocorticoids secretion (Cushing's Syndrome during active phase, treatment and under remission and newly or on established glucocorticoid replacement therapy adrenal insufficiency)

DETAILED DESCRIPTION:
This is an intervention, prospective, multicentric study.

Enrolled patients will undergo 4 visits:

* Adrenal insufficiency (AI) patients: patients affected by primary or secondary adrenal insufficiency, whether newly diagnosed or on established glucocorticoid therapy, will be evaluated at baseline and after one, three and six months.
* Cushing's Syndrome (CS) patients: patients affected by Cushing's Syndrome will be evaluated at baseline during active phase of the disease and one, three and six months after treatment or remission. Patients affected by Cushing's Syndrome who will require glucocorticoid replacement therapy after remission will be evaluated three and six months after remission and then three and six months after the eventual glucocorticoid replacement therapy withdrawal. CS treatment will be surgery or medical therapy according to guidelines. Timing of medical therapy administration will change during protocol according to circadian rhythms.

Age-, sex- and BMI- matched healthy controls will be enrolled. Patients and controls will undergo the same procedures at baseline and after 1, 3 and 6 months.

The primary outcome measure will be the evaluation of circadian genes CLOCK and Aryl Hydrocarbon Receptor Nuclear Translocator Like (ARNTL) expression in peripheral blood mononuclear cells (PBMC) compared to healthy controls.

Secondary Outcomes measures will be:

* Circadian genes expression assessment compared to healthy controls at 7:00-8:00 Ante Meridiem (AM) (before breakfast), 12:00 AM (before lunch), 3:00-4:00 Post Meridiem (PM) (after lunch), 7:00 PM (before dinner), 12:00 PM;
* Immune profiling compared to healthy controls by the quantification of peripheral blood mononuclear cells (PBMC) subpopulations assessed by flow cytometry at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM;
* Evaluation of inflammatory cytokines and adipokines production compared to healthy controls at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM;
* Circadian cortisol rhythm by serum and salivary dosage at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM;
* Sleep disturbances evaluation by The Pittsburgh Sleep Quality Index (PSQI) self reported questionnaire
* Evaluation of infectious diseases frequencies and severity compared to healthy controls. Infectious diseases will be evaluated by an adaptation of Infectious Diseases Questionnaire (GNC)
* Circadian blood pressure using ambulatory blood pressure monitoring blood pressure waves for a noninvasive estimation
* Quality of life using SF-36-Item Health Survey questionnaire
* Psychometric Evaluation using Beck Depression Inventory questionnaire
* Evaluation of sexual dysfunction using FSFI questionnaire in woman and IIEF questionnaire in man
* Evaluation of insuline resistance calculated with HOMA index
* Evaluation of body weight (kg)
* Evaluation of blood lipid profile

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary chronic adrenal insufficiency, previously or newly diagnosed.
* ACTH-dependent or ACTH-independent Cushing's Syndrome diagnosis during active disease (new diagnosis or recidivating).

  * Signed informed consent to participate in the study.

Exclusion Criteria:

- acute adrenal insufficiency;

* clinical or laboratory signs of significant respiratory, hepatobiliary, or pancreatic disease;
* pregnancy;
* severe infections, surgery, trauma requiring hospitalization within 3 months before study entry;
* any active blood or rheumatic disorders, and active liver disease in the previous 5 years;
* clinically significant chronic kidney disease;
* severe psychiatric diseases;
* history of neoplasms in the last 5 years (except for adrenal or pituitary adenoma in Cushing Syndrome, pituitary adenoma or related neolpasms in secondary adrenal insufficiency);
* heart disease with a class III or class IV functional capacity;
* BMI greater than 40 kg/m²;
* use of medication that interferes with cortisol metabolism within 1 month before study entry;
* treatment with systemic Glucocorticoid (GC) therapy other than hydrocortisone (HC), or cortisone acetate (CA);
* alcoholism and/or drug addictions;
* night-shift workers;
* use of melatonin, antipsychotic medications, estroprogestinic preparations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Circadian genes CLOCK and ARNTL expression evaluation | baseline, +1 month, +3 months, +6 months
  Change in relative expression circadian genes of CLOCK and ARNLT from baseline compared to healthy controls. After PBMC isolation by Ficoll-Plaque gradient, complementary DNA (cDNA) pool will be extracted and used as the template for subsequent Polymerase Chain Reaction (PCR) amplification in Real time PCR; Gene expression will be quantified as relative expression compared to housekeeping genes.

SECONDARY OUTCOMES:
Circadian gene expression profile | baseline, +1 month, +3 months, +6 months
  Change from baseline in relative expression and variations throughout the day of circadian genes (CLOCK and ARNTL) compared to healthy controls at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM. After PBMC isolation by Ficoll-Plaque gradient, cDNA pool will be extracted and used as the template for subsequent Polymerase Chain Reaction (PCR) amplification in Real time PCR; Gene expression will be quantified as relative expression compared to housekeeping genes.
Peripheral Blood Mononuclear Cells circadian profiling | baseline, +1 month, +3 months, +6 months
  Number of cells (number per mm3) of peripheral blood mononuclear cell subpopulations at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM
Circadian cortisol rhythm | baseline, +1 month, +3 months, +6 months
  Circadian cortisol rhythm by serum and salivary dosage at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM.
Sleep Disturbances | baseline, +1 month, +3 months, +6 months
  Sleep disturbances will be evaluated by The Pittsburgh Sleep Quality Index (PSQI). This questionnaire contains 19 self-related questions which are combined to create 7 component scores with a range of 0-3 points (0:no difficulty, 3: severe difficulty). Global score is the result to the addition of all component scores with a range of 0-21 points (0:no difficulty, 21: severe difficulty).
Infectious Diseases Frequency and Severity | baseline, +1 month, +3 months, +6 months
  Frequencies and severity of infectious diseases will be evaluated by modified Infectious Diseases Questionnaire (GNC).
  This questionnaire includes questions on infectious diseases of upper and lower respiratory tract, gastrointestinal tract, skin and urogenital tract contracted during the previous 12 months. Questions investigate on the number and duration of infections, necessity of antibiotic or antifungal therapy, hospital stay and days of absence from work. Final score represents the frequency of infections. Moreover, some questions investigate possible susceptible or protective factors for infectious diseases: vaccinations, use of corticosteroids, concomitant diseases, previous appendectomy, tonsillectomy, adenoidectomy, splenectomy or thymectomy.
Circadian blood pressure | baseline, +1 month, +3 months, +6 months
  Circadian blood pressure will be evaluated using ambulatory blood pressure monitoring blood pressure waves for a noninvasive estimation
Quality of life evaluation | baseline, +1 month, +3 months, +6 months
  Quality of life will be evaluated by the Physical Component score and the Mental Component score of the self-administered questionnaire SF-36-Item Health Survey questionnaire.
  This questionnaire measures eight scales: physical functioning, role physical, bodily pain, general health (physical component) and vitality, social functioning, role emotional, mental health (mental component).
  Interpretation of the score will be the following: at each item of the questionnaire corresponds a percentage value (from 0% to 100%). The average of the single items constitutes the scale total percentage (from 0% to 100%); missing data are not considered during calculation. High score defines a more favorable health state.
Psychometric Evaluation | baseline, +1 month, +3 months, +6 months
  Psychometric Evaluation will be evaluated using Beck Depression Inventory questionnaire. : a 21-item measure of depressive symptoms. Each answer is scored on a scale value (from 0 to 3 points). The global score is obtained adding all single scores, with a range of 0-63. Higher score constitutes worse burden of symptoms (0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression).
Sexual dysfunction in women | baseline, +1 month, +3 months, +6 months
  Evaluation of sexual dysfunction will be evaluated in women using FSFI questionnaire. This is a 19-item questionnaire that covers six domains: desire, arousal, lubrication, and orgasm, satisfaction, and pain. The ranges of the domain scores are as follows: for desire 1.2 - 6.0, for arousal, lubrication, orgasm and pain 0 - 6.0 and for satisfaction 0.8 - 6.0. The higher scores of the six domains indicate better sexual functioning about that domain. The overall FSFI score is obtained by summing the six domain scores. The overall FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
Sexual dysfunction in men | baseline, +1 month, +3 months, +6 months
  Evaluation of sexual dysfunction will be evaluated in men using IIEF questionnaire. The IIEF is an internationally validated test. It is used to assign a score of erectile dysfunction: severe score 1 to 10; moderate score 11 to 16; low to moderate score 17 to 21; Low score 22 to 25; no erectile dysfunction score 26 to 30
insuline resistance | baseline, +1 month, +3 months, +6 months
  Measurement of HOMA index calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
blood lipid profile | baseline, +1 month, +3 months, +6 months
  Measurement of Total Cholesterol, LDL cholesterol, HDL cholesterol, Triglyceredes
Inflammatory cytokines levels | baseline, +1 month, +3 months, +6 months
  Evaluation of Tumor Necrosis Factor alpha (TNFα), Transforming Growth Factor beta (TGF-β), Interferon gamma (IFN-γ), Leptin, Resistin, Adiponectin, Adipsin, Monocyte Chemoattractant Protein-1 (MCP-1), Serpin, C Reactive Protein (CRP), Interleukin 6 (IL-6), Interleukin 10 (IL-10) serum concentrations at 7:00-8:00 AM (before breakfast), 12:00 AM (before lunch), 3:00-4:00 PM (after lunch), 7:00 PM (before dinner), 12:00 PM

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Experimental Medicine, "Sapienza" University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided